CLINICAL TRIAL: NCT05060380
Title: Feasibility of a Novel Resistance Exercise in Individuals With Osteoporosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was never started.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Harshvardhan Singh, PRINCIPAL INVESTIGATOR, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 300004541
Record Dates: First submitted 2021-07-28; First posted 2021-09-29 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Osteopenia; Osteoporosis; Postmenopausal Osteoporosis; Sarcopenia
Keywords: aging; bone; muscle; exercise
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis; Osteoporosis, Postmenopausal; Sarcopenia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Individuals will be randomly assigned to exercise or no exercise group.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be blinded to the group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise training (Experimental): The exercise training group will receive progressive muscle resistive exercise, 10 sets of exercises for 2 times per week for a total of 6 months.
  Interventions: Other: Exercise training
- Control (No Intervention): The control group will be asked to maintain their normal lifestyle and will be advised to continue their standard care of treatment.

INTERVENTIONS:
Other: Exercise training — Progressive muscle resistive exercise will be performed by the experimental group only. Control group will maintain their normal level of daily activity.
  Arms: Exercise training

SUMMARY:
The aim of the 2 month randomized controlled trial is to investigate the feasibility of a novel progressive muscle resistance exercise in individuals with low bone mass.

DETAILED DESCRIPTION:
In 2008, medical cost of osteoporosis and osteoporosis-related fractures was estimated to be $22 billion. This is further expected to rise because of an increase of 20% in population with osteoporosis, amounting to 12 million adults over the age of 50 years, by 2020, out of which 80% will be postmenopausal women. Unfortunately, benefits due to pharmacological interventions have plateaued. Consequently, there is a critical need to identify complementary therapies to enhance the treatment of low bone mass in older adults. The aim of this study is to examine the feasibility of novel progressive muscle resistance exercise in postmenopausal women with low bone mass. Muscle will be assessed via imaging techniques and isokinetic dynamometer. Physical activity will be assessed via activity monitors. Blood will be collected to assess bone and muscle biomarkers. Balance will be assessed via clinical and biomechanical tests. Testing will be performed at 4 time points: baseline, 1 month, 3 month, and 6 months except imaging which will be done at the baseline and 6 months. The findings from this study will help us to understand the feasibility of resistive muscle exercise program in postmenopausal women with low bone mass.

ELIGIBILITY:
Inclusion Criteria:

* independent ambulatory
* diagnosed with low bone mass

Exclusion Criteria:

* uncontrolled hypertension
* secondary osteoporosis
* fragility fracture,
* clinical or laboratory evidence of hepatic
* renal disease,
* uncontrolled disorders of the parathyroid
* thyroid glands,
* a history of cancer in the past 5 years,
* any structured resistance training within the previous year, and
* past therapy with any drug for osteoporosis,
* any current therapy for osteoporosis except zoledronic acid,
* inability to walk independently or
* any other medical conditions which could restrict the potential participants from full participation as decided by their physician.

Ages: 55 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified as female.
Enrollment: 0 (Actual)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Bone biomarker | baseline
  bone formation and resorption marker
Bone biomarker | 1 month
  bone formation and resorption marker
Bone biomarker | 2 month
  bone formation and resorption marker

CONTACTS AND LOCATIONS:
Overall Officials: HARSHVARDHAN SINGH, PT, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No